CLINICAL TRIAL: NCT00103025
Title: Evaluation of the Mechanism of NO Formation and Pharmacokinetics of Long-Term Intravenous Nitrite Infusion in Healthy Volunteers
Brief Title: Nitrite Infusion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Russell R. Lonser, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050075; 05-N-0075
Record Dates: First submitted 2005-02-05; First posted 2005-02-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-10

CONDITIONS: Healthy
Keywords: Vasodilation; Hypotension; Hypertension; EDRF; Methemoglobinemia; Healthy Volunteer; HV
MeSH Terms: conditions — Aneurysm; Hypotension; Hypertension; Methemoglobinemia | interventions — Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite
Drug: Sodium Nitrite Injection

SUMMARY:
This study will determine the dose of sodium nitrite that can safely be used to prevent constriction, or tightening, of the arteries. Narrowed arteries in the brain can cause stroke. Animal studies show that nitrite injections improve blood flow and that injections over long periods of time prevent damage to the arteries in the brain; however, there is no information on the effects of prolonged nitrite infusion in humans. This study will establish the safe dose and side effects of nitrite infusion in humans.

Healthy normal volunteers between 21 and 60 years of age may be eligible for this study. Candidates are screened for high or low blood pressure, aspirin use, pregnancy, and blood levels of nitrite and methemoglobin (a substance that temporarily and slightly lowers the oxygen carried in the red blood cells). Pregnant women are excluded from the study.

Participants are admitted to the Clinical Center for 16 1/4 days, the first 2 days in the hospital's intensive care unit (ICU). Upon admission they provide a medical history, have physical and cardiovascular examinations, and blood tests. For the infusion procedure, a catheter (thin plastic tube) is inserted into an artery in the wrist or the crease of the elbow to measure blood pressure, and catheters are placed in a vein in each arm for administering the nitrite and withdrawing blood samples.

In the morning of day 1, after initial blood pressure and heart rate measurements are taken and a blood sample is drawn, a saline (salt water) infusion is started. Blood pressure and heart rate are monitored every 30 minutes for 6 hours, then every hour for 6 hours, then every 2 hours for 12 hours. Blood samples are collected every 4 hours for 24 hours. On day 2, the sodium nitrite infusion begins. Blood pressure and methemoglobin are monitored every 10 minutes for the first 2 hours. If blood pressure remains stable, the frequency of measurements is decreased to every 30 minutes for 4 hours, then every 1 hour for the next 6 hours, and then every 4 hours for 12 hours. If the pressure continues to remain stable, monitoring continues every 8 hours for the rest of the study. Blood is drawn periodically from the catheter to determine the amount of nitrite and methemoglobin in the body, with decreasing frequency from several times during the first hour of the infusion to every 24 hours. After the first 24 to 48 hours of the nitrite infusion, participants are transferred from the ICU to a general nursing unit fo...

DETAILED DESCRIPTION:
Nitric oxide (NO) is beneficial in treatment of many animal models of diseases like heart and brain ischemia, reperfusion injury, and delayed cerebral vasospasm after subarachnoid hemorrhage. It also has been shown to open blood-brain barrier facilitating transfer of chemotherapeutic agents, dilate constricted pulmonary arteries, and inhibit apoptosis, as well as modulate angiogenesis. Until recently, all these biological effects were attributed to the regional synthesis of nitric oxide by the endothelium and its local influence of vascular tone. However, "NO bioactivity" may be transported in blood and have biological effects at a distance from the site of entry into the circulation. These effects of NO are mediated by intravascular NO-stores. Candidates are protein and heme-bound NO species (RXNO) in plasma or erythrocytes and the oxidative NO-metabolite nitrite. Cumulating evidence suggests that nitrite may serve as a major intravascular storage pool for NO. Recent studies have shown that (1) regional, intra-arterial infusion of nitrite elicits a downstream vasodilator response in humans and (2) intravenous long-lasting administration prevents development of delayed cerebral vasospasm in a primate model of subarachnoid hemorrhage (SAH). These studies suggest a potential new therapeutic approach to many diseases. Despite extensive data documenting the pharmacokinetics and safety of the bolus and short intravascular infusions of nitrite, there are no human data evaluating safety and toxicity of prolonged delivery of nitrite, which would be required for treatment of vascular diseases.

OBJECTIVES

This study has the following objectives: (1) to determine the safety and (2) toxicity of a 48-hour and 14-day intravenous infusion of nitrite. The study should also help to elucidate the mechanism(s) through which nitrite ions contribute to vasodilation.

STUDY POPULATION

The study population will include sixteen 48-hour infusion healthy volunteers (out of 40 screened volunteers) of both genders, age 21-60, who will have a continuous intravenous infusion of sodium nitrite (the source of the drug will be determined by a CRADA).

DESIGN

This is a Phase I toxicity study of intermediate (48-hour) intravenous infusion of sodium nitrite in healthy volunteers.

OUTCOME MEASURES

Sixteen healthy volunteers of both genders, age 21-60, will have a 48-hour continuous intravenous infusion of sodium nitrite during which the subjects' clinical condition, blood levels of nitrite/methemoglobin, hematology, blood chemistry, and pressure will be meticulously monitored.

The first subject will receive the sodium nitrite infusion at 12 mg/48 hours. This dose, according to our knowledge from the former studies and detailed analysis of pharmacokinetics of sodium nitrite, will result in blood levels of sodium nitrite below 80 nmol/L, levels that are significantly below levels reported as normal (0.5 micromol/L to 1 micromol/L). Thus, we will use the modified accelerated titration design for Phase I Clinical studies. In the accelerated design the initial patient will start with the dose 1 nmol/min/kg/48hr, i.e. 12 mg total over 48 hours for a person weighting 60 kg. Cohorts of one new subject per dose level and double dose steps will be used during the initial accelerated stage. When the first instance of dose-limiting toxicity (DLT) is observed at any dose level, the next lower dose level cohort will be expanded to three patients and revert to the use of conventional modified Fibonacci escalation/de-escalation. If no DLT is observed at level 10, the cohort will be expanded to a total of three and de-escalated as appropriate. If no more than one subject among three patients experience DLT at this dose, level 10 will be considered to be the maximum tolerated dose (MTD).

The results of this 48-hour infusion phase 1 trial will be submitted to FDA before initiation of a 14-day clinical study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 21-60 years of age.

Subjects must be in good health.

Subjects must provide informed, written consent for participation in this study.

Female subjects of childbearing age must have a negative pregnancy test and agree to participate in assessment of menstrual cycle duration before, during, and after infusion.

Subjects must be willing to temporarily stop any medications (except oral contraception), vitamin supplements, herbal medicines.

Subjects will have hemoglobin levels above 11.1 g/dL.

EXCLUSION CRITERIA:

Subjects with a history or evidence of present or past hypertension (blood pressure greater than 140/90 mmHg), hypercholesterolemia (LDL cholesterol greater than 130 mg/dL), or diabetes mellitus (fasting blood glucose greater than 126 mg/dL).

Subjects who have a history of smoking within two years.

Subjects who have a history of cardiovascular disease, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

Subjects with red blood cell G6PD deficiency (levels below the lower limits of normal).

Subjects with a history of reaction to a medication or other substance characterized by dyspnea and cyanosis.

Subjects with a baseline methemoglobin level greater than 1%.

Pregnant women, since nitrite may cross the placenta; nitrite effect on fetus is unknown and mother's methemoglobinemia may be dangerous to the fetus.

Breast-feeding females, since nitrite crosses into breast milk and could cause methemoglobinemia in the infant.

Subjects with a blood pressure of less than 100/70 mmHg on the study day.

Subjects treated with nitrates (e.g. nitroglycerin).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-02-04; Primary Completion 2011-05-10 (Actual); Study Completion 2011-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Afshar JK, Pluta RM, Boock RJ, Thompson BG, Oldfield EH. Effect of intracarotid nitric oxide on primate cerebral vasospasm after subarachnoid hemorrhage. J Neurosurg. 1995 Jul;83(1):118-22. doi: 10.3171/jns.1995.83.1.0118. PMID 7782826
- [Background] Cosby K, Partovi KS, Crawford JH, Patel RP, Reiter CD, Martyr S, Yang BK, Waclawiw MA, Zalos G, Xu X, Huang KT, Shields H, Kim-Shapiro DB, Schechter AN, Cannon RO 3rd, Gladwin MT. Nitrite reduction to nitric oxide by deoxyhemoglobin vasodilates the human circulation. Nat Med. 2003 Dec;9(12):1498-505. doi: 10.1038/nm954. Epub 2003 Nov 2. PMID 14595407
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Derived] Pluta RM, Oldfield EH, Bakhtian KD, Fathi AR, Smith RK, Devroom HL, Nahavandi M, Woo S, Figg WD, Lonser RR. Safety and feasibility of long-term intravenous sodium nitrite infusion in healthy volunteers. PLoS One. 2011 Jan 10;6(1):e14504. doi: 10.1371/journal.pone.0014504. PMID 21249218